CLINICAL TRIAL: NCT04115111
Title: A Phase II Study to Investigate the Activity and Safety of Anti-PD-L1 Antibody (Durvalumab) In ADvancEd Pretreated Malignant Pleural Mesothelioma - DIADEM Study
Brief Title: Diadem to Investigate the Activity and Safety of Durvalumab
Acronym: Diadem
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRFMN-MPM-7109
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Pleura Mesothelioma
Keywords: malignant pleural mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab arm (Experimental): Patients will receive Durvalumab at the dose and regimens described above every 4 weeks until evidence of disease progression or occurrence of unacceptable toxicity.
  Patients who show evidence of disease progression but appear to tolerate Durvalumab well, for whom no other treatment options exist and who, at the judgement of the investigator, may still enjoy clinical benefit, will be classified as failures and offered the possibility to continue treatment with extended follow up.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab in monotherapy as second line treatment

SUMMARY:
Malignant pleural mesothelioma (MPM) is a cancer with high mortality rate and few therapeutic options.essentially all patients usually progress and die subsequently to a first line therapyl. There is strong evidence that the immune system is deeply involved in the biogenesis of MPM and that an imbalance in pro-inflammatory cytokines and exhausted adaptive T-cell mediated immune response are the main causes of neoangiogenesis, progression and metastatisation processes.Numerous Phase II-III clinical trials are underway evaluating Durvalumab either as monotherapy or combination with evidence of activity in a wide range of solid tumors. Durvalumab has received FDA approval as second line treatment in patients with locally advanced or metastatic urothelial carcinoma.

Given these prospects for PD-L1 Ab, a Phase II study is proposed in order to evaluate the activity and safety of Durvalumab in advanced pretreated MPM.

DETAILED DESCRIPTION:
Malignant pleural mesothelioma (MPM) is a cancer with high mortality rate and few therapeutic options. Its incidence is growing fast worldwide and is associated with asbestos exposure, a well known cancerogenic factor driving the development of this cancer. Generally MPM is diagnosed at an advanced inoperable stage and most frequently the only therapeutic approach is palliative chemotherapy. Platinum-pemetrexed doublets prolong significantly median overall survival (OS) and median progression free survival (PFS) with respect to platinum alone and are considered the only therapeutic option in a first line setting. Unfortunately, essentially all patients usually progress and die subsequently to a first line therapyl. There is strong evidence that the immune system is deeply involved in the biogenesis of MPM and that an imbalance in pro-inflammatory cytokines and exhausted adaptive T-cell mediated immune response are the main causes of neoangiogenesis, progression and metastatisation processes. Newer immunotherapeutic agents act on regulatory molecules expressed on immune cells in order to increase T cell activity and immune response against tumor. The anti-cytotoxic T lymphocyte antigen 4 (anti-CTLA4) demonstrated activity and a long-term disease control (DC) rate in advanced pretreated MPM in phase II study even if these results are not confirmed in more recently Phase IIb randomized trial versus placebo (DETERMINE study). Antibodies against Programmed Death 1 receptor (PD-1) and its ligand (PD-L1) are highly promising new agents regulating immune check-point processes. In particular the interaction of these agents takes place peripherally more than in the lymphoid tissue and may explain the higher response rate and lower adverse immune effects in comparison to antiCTLA4 agents. AntiPD-L1 antibodies are widely studied in many Phase I-II trials in different advanced pretreated solid tumors independent of tumor PD-L1 expression, with promising results and long-term survival. Ongoing melanoma and lung cancer phase III trials would probably better define the role of this class of drugs in clinical practice. Durvalumab is a human IgG1 antibody which binds specifically to PD-L1, preventing binding to PD-1 and CD80. Numerous Phase II-III clinical trials are underway evaluating Durvalumab either as monotherapy or combination with evidence of activity in a wide range of solid tumors. Durvalumab has received FDA approval as second line treatment in patients with locally advanced or metastatic urothelial carcinoma.

Given these prospects for PD-L1 Ab, a Phase II study is proposed in order to evaluate the activity and safety of Durvalumab in advanced pretreated MPM.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of advanced unresectable MPM;
2. Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (preferred) or at least 5 unstained slides for central determination of PD-L1 expression;
3. Aged ≥ 18 years;
4. Performance status 0-1 (ECOG);
5. Measurable disease as defined by Modified RECIST v1.1 for MPM;
6. One previous chemotherapy line for MPM, based on pemetrexed plus platinum derivative combination;
7. Previous chemotherapy course concluded at least 4 weeks prior to recruitment;
8. Signed informed consent;
9. Negative pregnancy test. All patients in reproductive age or potential must agree to use effective contraception, as defined by the study protocol for the entire duration of treatment with study drug and for 3 months following its interruption;
10. Patients who have received palliative radiation are eligible if <30% of bone marrow was irradiated and normal hematological function was completely regained;
11. Adequate organ and marrow function as defined below: Haemoglobin ≥ 9.0 g/dL, Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3), Platelet count ≥ 100 x 109/L (>100,000 per mm3);
12. Adequate liver function: Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (except for patients confirmed Gilbert's syndrome, who will be allowed only in consultation with their physician); AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN;
13. Adequate renal function: Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.

Exclusion Criteria:

1. Radiotherapy with curative intent to thoracic wall (concomitant with or prior to chemotherapy);
2. Severe concomitant illness;
3. History of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, type I diabetes mellitus, vasculitis, or glomerulonephritis;
4. Any other anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent);
5. History of primary immunodeficiency;
6. HIV( Ab anti HIV+), active TB infection , HBV or HCV infection;
7. History of allogeneic organ transplant;
8. History of hypersensitivity to durvalumab or any excipient;
9. Any condition that, in the opinion of the investigator, would interfere with study treatment or patient safety;
10. History of other malignancies (except basal cell carcinoma or cervical carcinoma in situ, adequately treated, melanoma stage one, prostate adenocarcinoma, bladder cancer), unless in remission for 3 years or more and judged of negligible potential of relapse;
11. Unstable cardiac condition, including congestive heart failure or angina pectoris, myocardial infarction within one year before enrolment, uncontrolled arterial hypertension or arrhythmias;
12. Brain / leptomeningeal involvement;
13. Any previous treatment with a PD-1 or PD-L1 inhibitor, including Durvalumab;
14. AEs from prior anticancer therapy that have not resolved to grade ≤ 1 except for alopecia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Proportion of survived patients at 16 weeks | 16 weeks
  Proportion of patients alive and free from progression or death at 16 weeks (PFS 16 w) calculated from the start of treatment (Durvalumab).

SECONDARY OUTCOMES:
Progression free survival | 16 weeks
  defined as the time from treatment start to progression of disease or death from any cause; in absence of an event, patients will be censored at the time of the latest date of assessment. If the patient has no evaluable visits or does not have baseline data they will be censored at 1 day.
overall survival | 16 weeks
  defined as the time from treatment start to death from any cause; in absence of an event, patients will be censored at the time of the latest date of assessment. If the patient has no evaluable visits or does not have baseline data they will be censored at 1 day.
Objective response rate | 16 weeks
  defined as the proportion of patients with complete response (CR) or partial response (PR) according to CT assessment using the RECIST v1.1 criteria modified for MPM (Modified RECIST). Independent central review will be used to confirm investigator ORR.
Tumour growth index | 16 weeks
  defined as the ratio between PFS and the time from treatment start to progression of disease in first-line treatment
Evidence of Number of Adverse Events | 16 weeks
  Evaluated based on frequency, type and severity of reported AEs, immune related irAE, clinical laboratory assessments, vital signs and physical examination. Adverse events will be encoded and graded using NCI-CTCAE version 4.03.
Exploratory endpoint | 16 weeks
  PD-L1 IHC expression in tumor samples and tumor infiltrating lymphocytes (TIL), measured with the validated ABCAM 28-8 assay IHC assay optimized for use on the automated BenchMark UTRA platform (Ventana Medical Systems, Tucson, AZ, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Diego Cortinovis, MD, Principal Investigator — ASST-Monza San Gerardo Hospital
Locations (1):
- San Gerardo Hospital, Monza, Italy

REFERENCES:
- [Result] Canova S, Ceresoli GL, Grosso F, Zucali PA, Gelsomino F, Pasello G, Mencoboni M, Rulli E, Galli F, De Simone I, Carlucci L, De Angelis A, Belletti M, Bonomi M, D'Aveni A, Perrino M, Bono F, Cortinovis DL; DIADEM groupD. Final results of DIADEM, a phase II study to investigate the efficacy and safety of durvalumab in advanced pretreated malignant pleural mesothelioma. ESMO Open. 2022 Dec;7(6):100644. doi: 10.1016/j.esmoop.2022.100644. Epub 2022 Dec 1. PMID 36463732